CLINICAL TRIAL: NCT03737591
Title: The Implication of Plasma Circulating Tumor DNA Methylation Haplotypes in Detecting Colorectal Cancer and Adenomas: a Multicenter, Cohort Study
Brief Title: The Implication of Plasma ctDNA Methylation Haplotypes in Detecting Colorectal Cancer and Adenomas
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Collaborators: Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Guoxiang Cai, Professor, Fudan University
Other Study IDs: FDCRCA-1
Record Dates: First submitted 2018-11-08; First posted 2018-11-09 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Colorectal Cancer; Adenoma
Keywords: Colorectal Cancer; Adenomas; ctDNA Methylation Haplotypes
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy individuals: Healthy individuals
  Interventions: Diagnostic Test: Next-generation sequencing (NGS)
- Patients with Colorectal cancer: Stage I-IV colorectal cancer patients
  Interventions: Diagnostic Test: Next-generation sequencing (NGS)
- Patients with Colorectal Adenomas: Patients with Colorectal Adenomas
  Interventions: Diagnostic Test: Next-generation sequencing (NGS)

INTERVENTIONS:
Diagnostic Test: Next-generation sequencing (NGS) — NGS test for colorectal tumor-specific plasma ctDNA methylation markers prior to endoscopy

SUMMARY:
This is a multicenter, clinical study. This study is to evaluate the sensitivity of plasma ctDNA methylation haplotypes in detecting colorectal cancer, adenoma and the specificity in healthy individuals.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common cancer worldwide, the second deadliest cancer in the United States. DNA methylation is a commonly used biomarker for non-invasive CRC detection in plasma. The low sensitivity of blood-based tests is due to several limitations of detecting ctDNA in early-stage cancer. We developed and validated a high-throughput methylation-based blood test highly sensitive for colorectal cancer and precancerous lesions. This previously established colorectal tumor-specific plasma ctDNA methylation markers (diagnostic model established by next-generation sequencing of gene loci methylation) had a high sensitivity in CRC patients and a high specificity in healthy individuals in a large retrospective sample study. This prospective, multicenter, clinical study is to further evaluate the sensitivity of plasma ctDNA methylation haplotypes in detecting colorectal cancer, adenoma and the specificity in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

Healthy Individuals:

* Written informed consent must be obtained from healthy individuals to comply with the requirements of the study.
* Healthy individuals who received colonoscopy.

Patients with Colorectal Cancer or Adenomas:

* Male or female ≥ 18 years of age on the day of signing informed consent.
* Patients need to receive surgical resection or endoscopic resection.
* Patients must have histologically confirmed stage I-IV colorectal cancer or adenomas
* Patients must have a performance status of ≤1 on the ECOG Performance Scale.
* Written informed consent must be obtained from patient or patient's legal representative and ability for patient to comply with the requirements of the study.

Exclusion Criteria:

* Patients received adjuvant treatment prior to the surgical resection.
* Patients received blood transfusion two weeks before or during the surgical resection.
* Patients with unresected advanced colorectal adenoma.
* Patients who are positive for Human Immunodeficiency Virus (HIV), Hepatitis B or Hepatitis C.
* Patients who are pregnant.
* Patients who are alcoholic or drug abusers.
* Patients with a history or current evidence of any condition or abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals and patients with stage I-IV colorectal cancer or adenomas must have baseline evaluations performed prior to the study and must meet all inclusion and exclusion criteria. In addition, the patient must be thoroughly informed about all aspects of the study, including the study visit schedule and required evaluations and all regulatory requirements for informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 1138 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity | 2 years
  The sensitivity of plasma ctDNA methylation haplotypes in detecting colorectal cancer and adenoma
Specificity | 2 years
  The specificity of plasma ctDNA methylation haplotypes in healthy individuals

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

REFERENCES:
- [Derived] Mo S, Dai W, Wang H, Lan X, Ma C, Su Z, Xiang W, Han L, Luo W, Zhang L, Wang R, Zhang Y, Zhang W, Yang L, Lu R, Guo L, Zheng Y, Huang M, Xu Y, Liang L, Cai S, Cai G. Early detection and prognosis prediction for colorectal cancer by circulating tumour DNA methylation haplotypes: A multicentre cohort study. EClinicalMedicine. 2022 Nov 3;55:101717. doi: 10.1016/j.eclinm.2022.101717. eCollection 2023 Jan. PMID 36386039